CLINICAL TRIAL: NCT04792710
Title: Randomised Trial Comparing Pre-operative Administration of Single Dose Kefazolin to Kefazolin Plus Metronidazole to Reduce Postpartum Infection
Brief Title: Kefazolin Versus Kefazolin Plus Metronidazole to Reduce Postpartum Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pretoria (Other)
Responsible Party: Principal Investigator, Leon Snyman, Prof, University of Pretoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PPS trial 1
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Prevention of Postpartum Sepsis
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Randomised placebo controlled trial
Who Masked: Outcomes Assessor
Masking Description: The out comes assessor will not have access to the arm the patient was randomised to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): This arm will be allocated to receive metronidazole 500 mg in addition to the current standard of care (Kefazolin 1 or 2 grams) administered intravenously prior to skin incision at caesarean section as a once off dose
  Interventions: Drug: Metronidazole
- Control arm (Placebo Comparator): This arm will be allocated to receive the current standard of care (Kefazolin 1 or 2 grams) administered intravenously prior to skin incision at caesarean section plus a placebo of normal saline 50 ml administered intravenously as a once off dose
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Metronidazole 500 mg intravenous stat dose prior to skin incision
  Other Names: Flagyl

SUMMARY:
Randomised controlled trial to investigate the efficacy of adding metronidazole pre-operatively to kefazolin in reducing postpartum infection

DETAILED DESCRIPTION:
All pregnant patients scheduled for emergency or elective Caesarean section ≥18 years, willing and able to provide informed consent and not receiving antibiotics, will be eligible for recruitment. Patients will be randomised into receiving kefazolin according to current standard of care administered pre-operatively intravenously with placebo (control arm), and kefazolin according to current standard of care administered pre-operatively with metronidazole 500 mg intravenously pre-operatively. Outcome measures will be surgical site infection, urinary tract infection and postpartum endometritis. Five hundred patients will be recruited in each arm

ELIGIBILITY:
Inclusion Criteria:

18 years and older Willing and able to provide written informed consent

Exclusion Criteria:

* women younger than 18 years women not able or willing to provide written informed consent women with or without infection already receiving antibiotics for other indications women allergic to kefazolin or metronidazole

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-08 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of reducing surgical site infection | Seven days post-operatively
  Incidence of surgical site infections

SECONDARY OUTCOMES:
Efficacy of reducing urinary tact infections | Three days post-operatively
  Incidence of urinary tract infections
Efficacy of reducing postpartum endometritis | Seven days post-operatively
  Incidence of endometritis

CONTACTS AND LOCATIONS:
Locations (1):
- Kalafong Provincial Tertiary Hospital, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No